CLINICAL TRIAL: NCT02355652
Title: Comparison of Two Surgical Strategies of Total Knee Arthroplasty : Cemented Versus Uncemented HLS Knee-Tec Prosthesis System. A Prospective Randomized Study.
Brief Title: Cemented Versus Uncemented Total Knee Arthroplasty : a Prospective Randomized Study
Acronym: HLS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: an other study will start with new outcome measures
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014.883
Record Dates: First submitted 2015-01-26; First posted 2015-02-04 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Total Knee Arthroplasty
Keywords: Total knee arthroplasty; IKS Score; cemented, uncemented

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cemented TKA (Active Comparator)
  Interventions: Device: Surgical total knee replacement using cemented components
- Uncemented TKA (Active Comparator)
  Interventions: Device: Surgical total knee replacement using uncemented components

INTERVENTIONS:
Device: Surgical total knee replacement using cemented components — Each patient of this arm will go under a surgical procedure of total knee replacement (or total knee arthroplasty) using cemented femoral and tibial prosthetic components.
  Arms: Cemented TKA
Device: Surgical total knee replacement using uncemented components — Each patient of this arm will go under a surgical procedure of total knee replacement (or total knee arthroplasty) using uncemented femoral and tibial prosthetic components.
  Arms: Uncemented TKA

SUMMARY:
The goal of this prospective randomized double-blind study is to compare clinical and radiological results of cemented and uncemented total knee arthroplasty (TKA).

Two hundred and fifty patients will be randomized in two groups : cemented TKA and uncemented TKA.

The primary outcome is the comparison of the International Knee Society (IKS) Score revised in 2011 at one year postoperative.

The second outcome is the comparison of standard one year-postoperative x-rays looking for signs of loosening.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis
* Need for a total knee arthroplasty

Exclusion Criteria:

* Age < 50 or > 80
* Need for a different procedure than a TKA
* Preoperative knee flexion < 90°
* Need for a TKA associated with a combined femoral or tibial osteotomy
* Knee already operated except for arthroscopy
* Mediocre bone quality

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
IKS 2011 Score measuring the clinical results of TKA | One year postoperative
  IKS 2011 Score will be assessed for each patients and the mean IKS Score will be compared between both arms

SECONDARY OUTCOMES:
Number of patients in each arm with radiological loosening signs of the TKA components | One year postoperative
  At one year postoperative, each patient will go under standard radiological exam seeking for signs of loosening of the prosthetic components. The number of patients presenting radiological signs of loosening will be compared between both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe NEYRET, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix-Rousse, Lyon, France

REFERENCES:
- See also: Related Info — http://www.orthopedie-lyon.fr